CLINICAL TRIAL: NCT02041819
Title: A Phase II Trial of Neoadjuvant Chemotherapy With Nimotuzumab Plus Nanoparticle Albumin-bound Paclitaxel and Cisplatin Followed by Surgery in Patients With Locally Advanced Squamous Cell Carcinoma of Esophagus
Brief Title: Neoadjuvant Chemotherapy of Nimotuzumab Plus Nab-Paclitaxel in Squamous Cell Carcinoma of Esophagus
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No recruitment
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Qiong Zhao, Chief of Department of Thoracic Oncology, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZYTOP1405
Record Dates: First submitted 2014-01-10; First posted 2014-01-22 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Squamous Cell Carcinoma of Esophagus
Keywords: Neoadjuvant chemotherapy; Nimotuzumab; Nab-Paclitaxel; Carcinoma of Esophagus
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma; Esophageal Neoplasms | interventions — nimotuzumab; Nimodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nimotuzumab nab-paclitaxel cisplatin (Experimental): Nimotuzumab: 200mg,IV once a week for 6 weeks during chemotherapy (days 1,8,15,22,29,36).
  Cisplatin: 75mg/m2,IV on days 1，22.
  Nab-paclitaxel: 125mg/m2,IV on days 1,8,22,29.
  patients will receive radical operation 4-6 weeks after Neoadjuvant therapy.
  Interventions: Drug: Nimotuzumab

INTERVENTIONS:
Drug: Nimotuzumab — Nimotuzumab: 200mg,IV once a week for 6 weeks during chemotherapy (days 1,8,15,22,29,36).
  Other Names: nimo

SUMMARY:
Nimotuzumab, a humanized monoclonal antibody against epidermal growth factor receptor (EGFR),has been shown to be effective and safe in some studies with head-neck cancers.Nab-paclitaxel regimen in advanced NSCLC has a better tumor response rate and safety than solvent-based paclitaxel.However,the safety and efficacy of Nimotuzumab plus nab-paclitaxel regimen is uncertain in neoadjuvant therapy in esophageal cancer.The investigators then initiated a phase II clinical trial with Nimotuzumab plus Nab-paclitaxel/cisplatin as the neoadjuvant chemotherapy in patients with locally advanced esophageal squamous cell carcinoma to observe the efficacy and safety of the combination.

DETAILED DESCRIPTION:
In the past decade, clinical trials have evaluated the role of neoadjuvant chemotherapy, radiation, or both, for patients with surgically resectable esophageal carcinoma, but have all failed to demonstrate a consistent survival benefit. In Eastern countries, preoperative chemotherapy followed by radical surgery became one of the treatment strategies for resectable, clinical stage II or III esophageal cancer. In an effort to improve the efficacy of systemic chemotherapy, we conducted a prospective study to evaluate the regimen of Nimotuzumab plus Nab-paclitaxel/cisplatin as perioperative therapy for patients with resectable esophageal squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed squamous cell carcinoma of the thoracic esophagus, including the gastroesophageal junction (Siewert type I)
* Locally advanced disease that is technically operable with curative intent (R0)
* T3, N0 OR T1-3, N+ OR T4, Nx
* No T1-2, N0
* No inoperable T4 (unequivocal organ involvement)
* No distant metastasis, including M1a lymph node status
* Lymph nodes suspicious of M1a status by CT scan, PET scan, or ultrasound must be verified by fine-needle aspiration cytology
* No carcinoma of the cervical esophagus
* Obstructive tumors allowed

Exclusion Criteria:

* Not suitable to surgery
* cervical Esophageal Carcinoma(distance of incisor tooth<19cm)
* early Esophageal Carcinoma(Stage I)
* complete esophageal obstruction，Esophageal perforation or hematemesis
* other malignant tumors, except for skin basal cell carcinoma, or cervical carcinoma in situ
* pregnant or breast-feeding women or people during the birth-period who refused to take contraceptives
* Uncontrolled seizures or psychiatric diseases, loss of control over their own behavior
* History of serious allergic or castor oil allergy
* Patients who are not suitable to participate in the trial according to researchers

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-02; Primary Completion 2016-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
response rate | From date of treatment until the date of progression, assessed up to 2 months
  pathological response rate and clinical response rate

SECONDARY OUTCOMES:
Overall survival | Overall survival was measured from the date of treatment to the date of death, or last follow-up,assessed up to 48 months
Progression-free survival | Progression-free survival was measured from the date of treatment to the date of first evidence of relapse or death due to any cause,assessed up to 36 months
Adverse events | During the chemotherapy,an expected average of 3 weeks
  Adverse events were classified according to U.S. National Cancer Institute common toxicity criteria, version 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Qiong Zhao, MD, Principal Investigator — The First Affiliated Hospital, Zhejiang University
Locations (1):
- The first affiliated hospital, Zhejiang University, Zhejiang, Zhejiang, China